CLINICAL TRIAL: NCT05466773
Title: Hemodialysis Eating Education Intervention to Improve the Depression, Treatment Adherence, Cardiovascular Risks, Quality of Life, and Healthcare Utilization Among Hemodialysis Patients: A Quasi-experimental Design
Brief Title: Hemodialysis Eating Education Intervention in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Taipei Medical University Hospital (Other); Cathay General Hospital (Other); Taipei Medical University WanFang Hospital (Other); Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Shwu-Huey Yang, Professor, Taipei Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TMU-JIRB：N201801034
Record Dates: First submitted 2022-07-14; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hemodialysis Complication
Keywords: hemodialysis, nutrition education

STUDY DESIGN:
Intervention Model Description: quasi-experimental design with 4 groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CN group (Experimental): Giving nutrition education for nurse, but not for patients
  Interventions: Behavioral: Hemodialysis eating index (HDEI) base education intervention
- CP group (Experimental): Giving nutrition education for patients, but not for nurses
  Interventions: Behavioral: Hemodialysis eating index (HDEI) base education intervention
- CNP group (Experimental): Giving nutrition education for both patients and nurses
  Interventions: Behavioral: Hemodialysis eating index (HDEI) base education intervention
- NC group (No Intervention): No nutrition education for patients and nurses

INTERVENTIONS:
Behavioral: Hemodialysis eating index (HDEI) base education intervention — The investigators have developed the educational materials for patients, in order to improve the dialysis outcomes. The interventions will be delivered to patients and nurses in hospital based hemodialysis centers.
  Arms: CN group; CNP group; CP group

SUMMARY:
The investigator aim to evaluate the effect of training program on treatment adherence, quality of life, cardiovascular risk factors, depression, and healthcare utilization. The investigator conducted a quasi experimental study. The investigator also examine the effect of interaction between health literacy and training program on depression, treatment adherence, cardiovascular risk factors, quality of life, and healthcare utilization.

The ultimate goal is to improve the dietary intake and dialysis outcomes for all hemodialysis patients in Taiwan. The investigator therefore will the SaaS dietary educational platform for this purpose.

DETAILED DESCRIPTION:
The investigator have completed the surveys on dietary intake, anthropometrics, clinical assessments, body compositions, and biochemical parameters and so on in designed hospitals. Assessment of cardiovascular disease risk factors: The diagnosed values were defined by the National Kidney Foundation Kidney Disease Outcomes Quality Initiative Work Group.

Health Literacy Health literacy will be also measured by Chew's 3 brief health literacy screening questions (BHLS), each with 5 possible response options [1]: (1) "How often do participants have problems learning about participants' medical condition because of difficulty understanding written information?" (always, often, sometimes, occasionally, or never); (2) "How often do participants have someone help participants read hospital materials?" (always, often, sometimes, occasionally, or never); and (3) "How confident are participants filling out medical forms by participants self?" (extremely, quite a bit, somewhat, a little bit, or not at all). The BHLS demonstrated evidence of construct validity among hemodialysis patients [2]. To identify the level of health literacy, sum scale of 3 screening questions will be calculate and classify into 3 levels: (1) Limited health literacy (=< 6 scale); (2) Marginal health literacy (7-8 scale); (3) Adequate health literacy (>= 9 scale) on the scale of 15 scale [3].

Dietary knowledge The dietary knowledge of nurses and patients will be evaluated pre-intervention and post-intervention, using a 10-item questionnaire developed by Kim and colleague [4]. The tool is to measure knowledge on protein, potassium, phosphorus, sodium, and water. The correct answer was treated as 'correct', incorrect or 'do not know' answers were treated as 'incorrect'; the highest scale possible was 10 points.

Treatment adherence Biological markers: The bio-markers to identify the dietary adherence are serum potassium (Pre-dialytic serum potassium ≤ 5.5 mEq/L), and phosphorus (Pre-dialytic serum phosphorus ≤ 4.5 mg/dL); fluid adherence is inter-dialysis weight gain (IDWG ≤ 4% of dry weight gain); medication adherence are (phosphate binders, antihypertensive, calcium supplements, and vitamin).

Self-report: The subjective adherence will be measured using the adherence behaviors subscale of the ESRD-Adherence Questionnaire (ESRD-AQ) [6]. The four subscales will be used which ask about treatment adherence to hemodialysis treatment (item 14 "During the last month, how many dialysis treatments did participants miss completely?", 17 "During the last month, how many times have participants shortened participants' dialysis time?", and 18 "During the last month, when participants' dialysis treatment was shortened, what was the average number of minutes?"), medications (item 26 "During the past week, how often have participants missed participants' prescribed medicines?"), fluid restrictions (item 31 "During the past week, how often have participants followed the fluid restriction recommendations?"), and diet recommendations (item 46 "During the past week, how many times have participants followed the diet recommendations?"). The ESRD-AQ is designed with the 5-point Likert scale, such that higher scales indicate better adherence.

Mental health The mental health was assessed by the Center for Epidemiologic Studies Short Depression Scale (CES-D 10). Patient will be asked about the ways they may have felt or behaved during the past week on the scale from rarely or none of the time to all of the time. Scale is the sum of the points for all 10 items. If more than 2 items are missing, do not scale. A scale of 10 or greater is considered depressed.

Quality of Life The quality of life among hemodialysis patients will be assessed using the Short Form-12 health survey subscale of the Kidney Disease and Quality of Life (KDQOL), with items measuring general health, activity limits (physical functioning), ability to accomplish desired tasks (role physical), role emotional, emotional well-being, energy level, pain, and social activities [7]. The SF-12 scale was validated in hemodialysis patients in Chinese population [8, 9].

Healthcare utilization Frequency of usage of emergency services, end-stage renal disease (ESRD)-related hospitalizations over past 6 months.

Patients' characteristics and health related behaviors Age (year), gender (male/female), marital status (married, single, divorce, widowed), highest education attainment (elementary school, junior high school, senior high school, college/university and above), ability to pay for medication (very difficult, fairly difficult, fairly easy, very easy), self-assessed social status (low, middle, high).

The physical activity was assessed by using valid and reliable Chinese version of the international physical activity questionnaire short form (IPAQ-SF) [10-12]. This 7-item survey aims to identify the frequency and duration of vigorous, moderate, and light PA, as well as inactivity during the past one week. Patients will be asked about frequency and amount of alcoholic beverage drinking in the last 30 days, and smoking status (non-smoker, occasional smoker, smoker).

ELIGIBILITY:
Inclusion Criteria:

Hemodialysis patients whose aged 20-75 years, received hemodialysis treatment thrice a week for at least 3 months, the education level of junior high school and higher, and Kt/V > 1.2.

Exclusion Criteria:

Hemodialysis patients with obvious edema, pregnancy, amputation, hyperthyroidism, hypothyroidism, malignancy, liver failure or cancer, mental disorders, tube feeding, hospitalization and plan to surgery, loss to measure body composition, and percentage body fat < 4% were excluded.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Health Literacy | baseline
  Health literacy will be also measured by Chew's 3 brief health literacy screening questions (BHLS), each with 5 possible response options: (1) "How often do you have problems learning about your medical condition because of difficulty understanding written information?" (always, often, sometimes, occasionally, or never); (2) "How often do you have someone help you read hospital materials?" (always, often, sometimes, occasionally, or never); and (3) "How confident are you filling out medical forms by yourself?" (extremely, quite a bit, somewhat, a little bit, or not at all).

SECONDARY OUTCOMES:
Dietary knowledge | 2 months
  The dietary knowledge of nurses and patients will be evaluated pre-intervention and post-intervention, using a 10-item questionnaire developed by Kim and colleague. The tool is to measure knowledge on protein, potassium, phosphorus, sodium, and water. The correct answer was treated as 'correct', incorrect or 'do not know' answers were treated as 'incorrect'; the highest scale possible was 10 points.

OTHER OUTCOMES:
Treatment adherence-biological markers | 4 months
  Biological markers: serum potassium, and phosphorus; inter-dialysis weight gain.
  Self-report: hemodialysis treatment, "During the last month, how many times have you shortened your dialysis time?", and "During the last month, when your dialysis treatment was shortened, what was the average number of minutes?"), medications, fluid restrictions, and diet recommendations
Treatment adherence-hemodialysis treatment | 4 months
  Hemodialysis treatment, "During the last month, how many times have you shortened your dialysis time?"
Mental health | 4 months
  The mental health was assessed by the Center for Epidemiologic Studies Short Depression Scale (CES-D 10).
Patients' characteristics and health related behaviors | baseline
  Age (year), gender (male/female), marital status (married, single, divorce, widowed), highest education attainment (elementary school, junior high school, senior high school, college/university and above), ability to pay for medication (very difficult, fairly difficult, fairly easy, very easy), self-assessed social status (low, middle, high).
  The physical activity was assessed by using valid and reliable Chinese version of the international physical activity questionnaire short form (IPAQ-SF). This 7-item survey aims to identify the frequency and duration of vigorous, moderate, and light PA, as well as inactivity during the past one week. Patients will be asked about frequency and amount of alcoholic beverage drinking in the last 30 days, and smoking status (non-smoker, occasional smoker, smoker).
Healthcare utilization | 4 months
  Frequency of usage of emergency services, end-stage renal disease (ESRD)-related hospitalizations over past 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Shwu-Huey Yang, Ph.D, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Other (Non U.s.), Taiwan

IPD SHARING:
Plan to Share IPD: No
We need more time to clear the data.

REFERENCES:
- [Background] Chew LD, Bradley KA, Boyko EJ. Brief questions to identify patients with inadequate health literacy. Fam Med. 2004 Sep;36(8):588-94. PMID 15343421
- [Background] Cavanaugh KL, Osborn CY, Tentori F, Rothman RL, Ikizler TA, Wallston KA. Performance of a brief survey to assess health literacy in patients receiving hemodialysis. Clin Kidney J. 2015 Aug;8(4):462-8. doi: 10.1093/ckj/sfv037. Epub 2015 Jun 10. PMID 26251719
- [Background] Wallace LS, Rogers ES, Roskos SE, Holiday DB, Weiss BD. Brief report: screening items to identify patients with limited health literacy skills. J Gen Intern Med. 2006 Aug;21(8):874-7. doi: 10.1111/j.1525-1497.2006.00532.x. PMID 16881950
- [Background] Duff EA, Chawke FM. A service review to assess if innovative intensive phosphate dietary education can help reduce phosphate levels to the recommended range in a hemodialysis population. Hemodial Int. 2017 Oct;21 Suppl 2:S22-S26. doi: 10.1111/hdi.12593. PMID 29064180
- [Background] Kim Y, Evangelista LS, Phillips LR, Pavlish C, Kopple JD. The End-Stage Renal Disease Adherence Questionnaire (ESRD-AQ): testing the psychometric properties in patients receiving in-center hemodialysis. Nephrol Nurs J. 2010 Jul-Aug;37(4):377-93. PMID 20830945
- [Background] Hays RD, Kallich JD, Mapes DL, Coons SJ, Carter WB. Development of the kidney disease quality of life (KDQOL) instrument. Qual Life Res. 1994 Oct;3(5):329-38. doi: 10.1007/BF00451725. PMID 7841967
- [Background] Wan EY, Chen JY, Choi EP, Wong CK, Chan AK, Chan KH, Lam CL. Patterns of health-related quality of life and associated factors in Chinese patients undergoing haemodialysis. Health Qual Life Outcomes. 2015 Jul 29;13:108. doi: 10.1186/s12955-015-0308-3. PMID 26215978
- [Background] Joshi VD, Mooppil N, Lim JF. Validation of the kidney disease quality of life-short form: a cross-sectional study of a dialysis-targeted health measure in Singapore. BMC Nephrol. 2010 Dec 20;11:36. doi: 10.1186/1471-2369-11-36. PMID 21172008
- [Background] Macfarlane DJ, Lee CC, Ho EY, Chan KL, Chan DT. Reliability and validity of the Chinese version of IPAQ (short, last 7 days). J Sci Med Sport. 2007 Feb;10(1):45-51. doi: 10.1016/j.jsams.2006.05.003. Epub 2006 Jun 30. PMID 16807105
- [Background] Liou YM, Jwo CJ, Yao KG, Chiang LC, Huang LH. Selection of appropriate Chinese terms to represent intensity and types of physical activity terms for use in the Taiwan version of IPAQ. J Nurs Res. 2008 Dec;16(4):252-63. doi: 10.1097/01.jnr.0000387313.20386.0a. PMID 19061172